CLINICAL TRIAL: NCT06575920
Title: Breathing Therapy for Patients With Medically Unexplained Physical Symptoms and Dysfunctional Breathing: A Pilot and Feasibility Study
Brief Title: Breathing Therapy for Patients in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Agder (Other)
Collaborators: UiT The Arctic University of Norway (Other); The University of New South Wales (Other)
Responsible Party: Principal Investigator, Tor Ivar Karlsen, Professor, University of Agder
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UAgder
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Mind-Body Therapies

STUDY DESIGN:
Intervention Model Description: Pilot and fesability study.
Masking Description: The principal investigator kept all records and collected data, which was blinded from the care provider, whose role was solely to perform lectures and exercises.,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients who met the inclusion criteria were asked by the GP if they wanted to participate in the study and, if accepted, their contact information was sent to the researchers (N=18). At the first session, the researcher informed participants of the content and duration of the intervention programme and collected signed informed consent from a total of 15 participants.
  Interventions: Behavioral: Breathing excercizes

INTERVENTIONS:
Behavioral: Breathing excercizes — The intervention comprised six sessions. The first week involved obtaining informed consent, taking measurements and providing a brief introduction to breath and coherent breathing exercises. This was followed by four weekly sessions, each consisting of 90 minutes combining lectures and breathing exercises. At the final session, measurements and feasibility data were collected.

SUMMARY:
Medically unexplained physical symptoms (MUPS) capture conditions characterized by symptoms without corresponding objective findings, such as asthenia, low back pain, fibromyalgia, irritable bowel syndrome, or chronic fatigue syndrome. In order to establish the grounds for a RCT. this pilot study aims to investigate the effectiveness and feasibility of a 5-week breathing retraining programme on patients who meet the criteria for MUPS.

DETAILED DESCRIPTION:
Medically unexplained physical symptoms (MUPS) are symptoms without an identifiable organic cause that lead to functional impairment. MUPS is highly prevalent in general practice consultations. This pilot study aimed to investigate the effectiveness and feasibility of a 5-week breathing retraining program for patients meeting the criteria for MUPS. The study used a quantitative observational design with pre- and post-intervention measurements. Fifteen participants with MUPS and dysfunctional breathing (assessed by the Nijmegen Questionnaire) were recruited from two general practitioner offices. The intervention consisted of 5 weekly sessions including education on breathing physiology and weekly breathing exercises focused on nasal breathing and resonance breathing techniques. One week post intervention, improvements were observed in dysfunctional breathing scores, lower symptom severity, higher general well-being, and reduced musculoskeletal pain complaints. At 3 months post-intervention, sustained improvements were seen in dysfunctional breathing, general well-being, musculoskeletal pain, and additionally lower pseudoneurological, gastrointestinal, and allergy complaints, as well as lower overall symptom burden and improved end-tidal CO2 levels.

The study concluded that the 5-week breathing program showed promising results for improving multiple patient-reported outcomes in MUPS. Recruitment, adherence, and acceptability of the program were satisfactory. A randomized controlled trial is recommended to further evaluate the efficacy of this breathing intervention for MUPS patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* dysfunctional breathing,
* sufficient laguage skills to fill out forms

Exclusion Criteria:

* Participants with asthma
* Participants with,chronic obstructive pulmonary disease
* Participants with respiratory allergy that is not optimally treated medically.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Nijmegen Questionnaire | Base line, end of intervention, and 3 months post-interventions
  To detect dysfunctional breathing (DB). The NQ consists of 16 questions ranked on a five-point Likert scale where "never" counts as 0 and "very often" counts as 4, giving a total DB score between 0-64. Healthy, asymptomatic individuals generally have a DB score between 7-12. A score above 19 is suggestive of DB.
Subjective Health Complaints Inventory | Base line, end of intervention, and 3 months post-interventions
  Measures 29 subjective health problems. The form lists 29 common somatic and psychological ailments, where the degree of complaints and duration must be stated for the last 30 days, graded on a four-point scale. The 29 individual health issues were grouped into five sub-issues [musculoskeletal pain (8 items), pseudoneurology (7 items), gastrointestinal disorders (7 items), allergic disorders (5 items), colds (2 items)], and a total score comprising all items. All scales were scored 0-100 (where 0 indicates no symptom pressure and 100 the highest possible symptom pressure).
Measure Yourself Medical Outcome Profile | Base line, end of intervention, and 3 months post-interventions
  Participants are asked to rate four items (symptom 1, symptom 2, well-being, and impact of symptoms on their daily activity status) on a scale of 0-6 where 0 is "As good as it could be" and 6 is "As bad as it could be". Participants report one or two symptoms (physical or mental) which bother them the most, consider how bad each symptom was during the last week, and score them accordingly. They also report how much these symptoms affected a particular activity, their well-being during the last week, use of medication, and any possible adverse effects or worsening of symptoms. The symptom pressure and general well-being (scales 0-6) are presented.
Carbon dioxide levels | Base line, end of intervention, and 3 months post-interventions
  End-tidal CO2 (EtCO2) (Microstream™) is an objective measure of hyperventilation and is easily detected through a nasal cannula with a capnograph together with respiratory rate (RR). The normal values of EtCO2 are 4.7 kPa - 6 kPa (45). Values below 4.6 are regarded as hypocapnia.
Heart rate variability | Base line, end of intervention, and 3 months post-interventions
  The registrations of HRV were performed using HeartMath with the participants in a sitting position, relaxed, and breathing regularly. In the 1990s, HeartMath Institute researchers identified a physiological state called heart coherence. Physiologically, the coherence state is marked by the development of a smooth, sine-wave-like pattern in the heart rate variability trace. This characteristic pattern, called heart rhythm coherence, is the primary indicator of the psychophysiological coherence state. The emWave Coherence score is a measure of the degree of coherence in the heart rhythm pattern. A coherent heart rhythm is a stable, regular, repeating rhythm resembling a sine wave at a single frequency between 0.04 - 0.24 Hz (3 - 15 cycles per minute). The more stable and regular the heart rhythm frequency, the higher the coherence score. Scores range from 0 - 16.

SECONDARY OUTCOMES:
Patient adherence and attrition rates | Base line, end of intervention, and 3 months post-interventions
  Number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Silje Haugland, PhD, Study Director — University of Agder
Locations (1):
- University of Agder, Arendal, Agder, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data presented in the published paper will be available to other researchers.
Time Frame: The data will be available after acceptance from a scientific journal for a period of five years.
Access Criteria: Data will be deposited at Sikt - Norwegian Agency for Shared Services in Education and Research
URL: https://sikt.no/

REFERENCES:
- [Derived] Svenningsen H, Stub T, Courtney R, Karlsen TI. Breathing therapy for patients with medically unexplained physical symptoms and dysfunctional breathing: A pilot and feasibility trial. PLoS One. 2025 Jul 11;20(7):e0325951. doi: 10.1371/journal.pone.0325951. eCollection 2025. PMID 40644391